CLINICAL TRIAL: NCT00603915
Title: Phase II Trial of Gemcitabine and Cisplatin/Carboplatin (GC) Plus Erlotinib in Patients With Recurrent and/or Metastatic Nasopharyngeal Cancer
Brief Title: A Study of Gemcitabine and Cisplatin/Carboplatin Plus Erlotinib in Patients With Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-774; NPC-774
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Nasopharyngeal Cancer
Keywords: gemcitabine; carboplatin; cisplatin; erlotinib; tarceva; nasopharyngeal
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Gemcitabine; Carboplatin; Cisplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GC Plus Erlotinib (Experimental): Eligible patients are treated with cisplatin/carboplatin and gemcitabine (GC) for 6 cycles of therapy followed by maintenance erlotinib. Those patients achieving SD or PR with chemotherapy will be started on maintenance erlotinib until disease progression. Those patients achieving CR with chemotherapy will be started on erlotinib for 6 cycles of treatment and those achieving CR on erlotinib will be treated with a maximum of 6 further cycles of erlotinib. Those patients with disease progression while on chemotherapy will be offered erlotinib 2 weeks following the last dose of chemotherapy until further disease progression.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin/Cisplatin; Drug: erlotinib

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m^2 intravenous (IV) day 1 and day 8
Drug: Carboplatin/Cisplatin — Area under curve (AUC)=5 (Carboplatin) or 70mg/m^2 (Cisplatin) intravenous (IV) day 1
Drug: erlotinib — 150mg daily (post GC therapy)

SUMMARY:
Cisplatin or Carboplatin will be given on day 1 every 21 days for 6 cycles; Gemcitabine will be given on day 1 and day 8 every 21 days for 6 cycles. Those patients that do not progress on GC after 6 cycles of chemotherapy will be started on erlotinib daily until disease progression. A cycle of erlotinib will be 28 days. Patients who progress on GC will be offered erlotinib as well,in order to evaluate its activity as a single-agent in the second-line setting.

Patients previously treated with GC have reported a progression-free survival (PFS) of 9 months. We would anticipate an extension of PFS to 12 months in patients treated with GC followed by maintenance erlotinib. Furthermore, we hypothesize that patients who achieved benefit from GC therapy would have further response when treated with maintenance erlotinib, such that this strategy may increase the likelihood of attaining long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed World Health Organization (WHO) type I (keratinizing squamous cell carcinoma) or WHO type II a or b (differentiated non-keratinizing carcinoma or undifferentiated carcinoma) NPC.
* Presence of clinically and/or radiologically documented disease. At least one site of disease must be unidimensionally measurable as follows:

  * X-ray, physical exam > 20 mm
  * Spiral CT scan > 10 mm
  * Non-spiral CT scan > 20 mm
* Investigations including chest x-ray or CT scan of chest, CT or MRI of head and neck (for patients with locally advanced or locally recurrent disease) and other scans as necessary to document all sites of study disease have been performed within 28 days prior to randomization. (Exceptions will be made only for patients who have negative examinations within 35 days prior to registration; exceptions for bone scans will be made for negative examinations within 60 days prior to registration.)
* Age > 18 years.
* ECOG performance status of 0,1 or 2 (see Appendix II).
* Patients must have a life expectancy of at least 12 weeks.
* Previous Therapy:

  * Chemotherapy: Advanced Disease: Patients may not have had prior therapy for recurrent or metastatic disease.
  * Curative Therapy: Patients may have had prior chemotherapy (including cisplatin/ carboplatin based regimens) in the neoadjuvant, concurrent and adjuvant setting for locally advanced nasopharyngeal carcinoma provided that 4 weeks have elapsed since treatment and any residual treatment related neuropathy or ototoxicity is < grade 1 for cisplatin dosing on this trial. Patient with neuropathy or ototoxicity > grade 2 will be dosed with carboplatin if otherwise eligible for this trial.
  * Radiation: Patients may have received prior radiotherapy provided that the last fraction was given at least 4 weeks prior to registration and all toxicities have resolved. If radiotherapy was delivered to the only site of measurable disease, then progression must have been documented in that site after completion of radiotherapy and prior to registration.
  * Previous Surgery: Previous major surgery is permitted provided that it has been at least 21 days prior to patient registration and that wound healing has occurred.
* Laboratory Requirements (must be done within 7 days prior to registration)

  * Hematology:

    * granulocytes (AGC) > 1.5 x 109/L
    * platelets > 100 x 109/L
  * Chemistry:

    * AST < 2.5 x UNL
    * ALT < 2.5 x UNL
    * Creatinine clearance(*) : CrCl > 60mls/min for cisplatin or CrCl between 30 - 59ml/min for Carboplatin

(*) calculated

* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. The patient must sign the consent form prior to randomization or registration.
* Patients must be accessible for treatment and follow up.
* Normal serum calcium

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 5 years.
* Patients with non-measurable disease only. (Please note that bone metastases are considered non-measurable).
* Pregnant or lactating women. However, if the patient is of childbearing potential, a urine β-HCG must be proved negative within 7 days prior to registration. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
* Patients with known brain metastases. (A head CT is not necessary to rule out brain metastases, unless there is clinical suspicion of CNS involvement).
* Serious illness or medical condition, which would not permit the patient to be managed according to the protocol including, but not limited to:
* History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements;
* Active uncontrolled infection;
* Symptomatic congestive heart failure, unstable angina, cardiac arrhythmia.
* Prior anti-EGFR monoclonal antibody or tyrosine kinase inhibitors.
* Any inflammatory changes of the surface of the eye.
* Hypersensitivity to erlotinib (Tarceva) or to any of the excipients
* Concomitant requirement for medications classified as CYP3A4 inducer or inhibitor. Inhibitors of CYP3A4 are prohibited beginning at least seven (7) days prior to the administration of the first dose of study medication and for the duration of the study. Inducers of CYP3A4 are prohibited beginning at least fourteen (14) days prior to the administration of the first dose of study medication and for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] You B, Le Tourneau C, Chen EX, Wang L, Jarvi A, Bharadwaj RR, Kamel-Reid S, Perez-Ordonez B, Mann V, Siu LL. A Phase II trial of erlotinib as maintenance treatment after gemcitabine plus platinum-based chemotherapy in patients with recurrent and/or metastatic nasopharyngeal carcinoma. Am J Clin Oncol. 2012 Jun;35(3):255-60. doi: 10.1097/COC.0b013e31820dbdcc. PMID 21358293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was activated on 14-June-2006. Patients with nasopharyngeal carcinoma meeting the eligibility criteria specified in the protocol were enrolled.
Groups:
- GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB: patients with recurrent and/or metastatic NPC will be treated with 6 cycles of GC followed by maintenance erlotinib (150mg by mouth daily) for 6 cycles.
Period: Overall Study
Arm/Group | GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB
Started | 20
Completed | 19
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  Canada | 20
Performance Status [Number; unit: Participants] — ECOG Performance Status is a scale and criteria to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. A lower ECOG indicates a better outcome.
  0 - fully active
  1. - restricted in physically strenuous activity
  2. - able to do selfcare, but unable to carry out any work activities
  3. - capable of only limited selfcare
  4. - completely disabled
  5. - dead
  Participants
    0 | 10
    1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival.
Description: From randomization to the first documented disease progression or death from any cause, whichever came first, assessed until all participants randomized to the study have progressed for died.
Time Frame: From the on-study date until the date of first documented progression or date of death from any cause any cause until all participants have progressed or died.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB
Number analyzed (Participants) | 19
Months | 6.3 [5.0 to 8.6]

2. Secondary Outcome: Number of Participants With the Responses Outlined
Description: Complete Response (CR): disappearance of all clinical and radiological evidence of tumour.
  Partial Response (PR): at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  Progressive Disease (PD): at least a 20% increase in the sum of LD of measured lesions taking as references the smallest sum LD recorded since the treatment started. Appearance of new lesions will also constitute progressive disease.
Time Frame: Measured every 2 cycles until the participant is off treatment.
Measure: Number; unit: Participants
Arm/Group | GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB
Number analyzed (Participants) | 19
Participants
  Complete Response | 0
  Partial Response | 7
  Stable Disease | 11
  Progressive Disease | 1
  Inevaluable | 1

ADVERSE EVENTS:
Arm/Group | GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB (N=20)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (3)
Stroke (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEMCITABINE AND CISPLATIN/CARBOPLATIN (GC) PLUS ERLOTINIB (N=20)
Hemoglobin decreased (Blood and lymphatic system disorders) | 19 (19)
Lymphocyte Count decreased (Blood and lymphatic system disorders) | 19 (19)
Leukocyte count decreased (Blood and lymphatic system disorders) | 18 (19)
Fatigue (General disorders) | 17 (17)
Neutrophil count decreased (Blood and lymphatic system disorders) | 18 (18)
Pain (General disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No